CLINICAL TRIAL: NCT01317524
Title: The Effects of Homogenized and Unhomogenized Milk on Postprandial Metabolism in Healthy Overweight Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Dairy Association (NZO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MEC 10-3-089
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Hyperlipidemias; Inflammation; Atherosclerosis
Keywords: Milk; Homogenization; Postprandial hyperlipidemia; Postprandial inflammation; Overweight
MeSH Terms: conditions — Hyperlipidemias; Inflammation; Atherosclerosis; Overweight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Homogenized Milk (Experimental): 900 mL homogenized milk is consumed within a mixed meal
  Interventions: Dietary Supplement: Homogenized milk
- Unhomogenized Milk (Experimental): 900 mL unhomogenized milk is consumed within a mixed meal
  Interventions: Dietary Supplement: Unhomogenized milk
- Skimmed Milk (Experimental): 900 mL skimmed milk and 44 g of butter are consumed within a mixed meal
  Interventions: Dietary Supplement: Skimmed Milk

INTERVENTIONS:
Dietary Supplement: Homogenized milk — 900 mL homogenized milk 2 slices of bread with marmalade 2 pieces of crisp bread
  Arms: Homogenized Milk
Dietary Supplement: Unhomogenized milk — 900 mL unhomogenized milk 2 slices of bread with marmalade 2 pieces of crisp bread
  Arms: Unhomogenized Milk
Dietary Supplement: Skimmed Milk — 900 mL skimmed milk 44 g of salted butter 2 slices of bread 2 pieces of crisp bread
  Arms: Skimmed Milk

SUMMARY:
The purpose of this study is to compare the effects of homogenized, unhomogenized and skimmed milk on postprandial metabolism in healthy overweight men

ELIGIBILITY:
Inclusion Criteria:

* men
* aged between 18 and 70 years
* Quetelet index between 25 - 30 kg/m2
* mean serum triacylglycerol (≤1.7 mmol/L (31))

Exclusion Criteria:

* women
* indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus (32)
* lactose intolerance
* current smoker
* familial hypercholesterolemia
* abuse of drugs
* more than 21 alcoholic consumptions per week
* no stable body weight (weight gain or loss < 3 kg in the past three months)
* use of medication or a diet known to affect serum lipid or glucose metabolism
* severe medical conditions that might interfere with the study, such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel diseases and rheumatoid arthritis.
* active cardiovascular disease like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebro vascular accident)
* use of an investigational product within the previous 1 month
* not willing to stop the consumption of vitamin supplements, fish oil capsules or products rich in plant stanol or sterol esters 3 weeks before the start of the study
* not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study
* difficult venipuncture as evidenced during the screening visits

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incremental Area Under the triacylglycerol Curve | during 8 hours after meal consumption

SECONDARY OUTCOMES:
Plasma inflammatory markers | during 8 hours after meal consumption
Markers of endothelial activation | during 8 hours after meal consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands